CLINICAL TRIAL: NCT00743717
Title: Clinical Trial on the Zirconia Femoral Component for the Gem Total Knee System
Brief Title: Evaluation of the Safety and Effectiveness of the Kinamed Gem Ceramic Femoral Component for Total Knee Replacement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kinamed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: G010204
Record Dates: First submitted 2008-08-27; First posted 2008-08-29 (Estimated); Results first posted 2013-05-22 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Knee Osteoarthritis
Keywords: total knee arthroplasty; osteoarthritis; ceramic bearing; zirconia
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Device: zirconia femoral component
- 2 (Active Comparator)
  Interventions: Device: cobalt chrome femoral component

INTERVENTIONS:
Device: zirconia femoral component — total knee arthroplasty performed using implant with zirconia femoral component
  Arms: 1
Device: cobalt chrome femoral component — total knee arthroplasty performed using implant with cobalt chrome femoral component
  Arms: 2

SUMMARY:
The aim of this study is to provide evidence that the safety and effectiveness of the ceramic femoral component of the Gem Total Knee System is similar to FDA approved implants used in total knee replacement surgery. The hypotheses to be tested are that the investigational and control groups are equivalent in terms of patient success rate and complication-free rate.

DETAILED DESCRIPTION:
Due to excellent biocompatibility and wear characteristics, ceramics have a long history of success in total hip arthroplasty (THA). Use of a ceramic-polyethylene wear couple in total knee arthroplasty (TKA) has shown promising laboratory and early clinical results. The use of ceramics in this study is intended to address long-term failure of TKA due to osteolysis associated with polyethylene wear debris.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature
* Primary TKA for osteoarthritis or post-traumatic arthritis of the knee joint
* Stable or reconstructable collateral and posterior cruciate ligaments
* Correctable deformity
* Intact quadriceps and hamstrings mechanisms
* Patella bone thick enough (at least 15 mm) after resection

Exclusion Criteria:

* Previous TKA
* Bilateral knee arthritis
* Non-availability for follow-up
* Mental incompetence or confinement
* Patients being treated with other investigational devices for same disorder
* Infection
* Osteoporosis, acute renal failure, or other disorders known to affect bone quality
* Charcot's or Paget's disease
* Patient physical condition preventing use of appropriate size implant
* Disease conditions affecting blood supply to knee
* Insufficient bone quality or quantity
* Physical condition predisposing implant to extreme loads
* History of septic knee arthritis
* History of drug abuse

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2004-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vineet Sarin, PhD, Study Director — Kinamed Incorporated

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited during pre-op TKA clinical exam during year 2004.
Groups:
- 1: Zirconia Femoral: zirconia femoral component : total knee arthroplasty performed using implant with zirconia femoral component
- 2: CoCr Femoral: cobalt chrome femoral component : total knee arthroplasty performed using implant with cobalt chrome femoral component
Period: Overall Study
Arm/Group | 1: Zirconia Femoral | 2: CoCr Femoral
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1: Zirconia Femoral | 2: CoCr Femoral | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 1 | 2 | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 62.5 (13.4) | 65.5 (4.94) | 64 (8.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Knee Score at 2 Years Post Operation
Description: The criterion used to assess the outcome is a Knee Score (as defined by Knee Society Clinical Rating System) > 80 points at two-years follow-up. This scoring system is defined in the following paper: Insall JN, Dorr LD, Scott RD, and Scott WN (1989). Rationale of the Knee Society clinical rating system. Clin Orthop(248): 13-4. The scale ranges from minimum of 0 (worst) to maximum of 100 (best). Knee Score > 80 was used as a criterion to assess "success".
Time Frame: within 2 years
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | 1: Zirconia Femoral | 2: CoCr Femoral
Number analyzed (Participants) | 2 | 2
units on a scale | 91 [85 to 97] | 89 [88 to 90]

ADVERSE EVENTS:
Arm/Group | 1: Zirconia Femoral | 2: CoCr Femoral
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No